CLINICAL TRIAL: NCT03982849
Title: Comparison of Topical Silymarin With Hydroquinone in the Treatment of Melasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Principal Investigator, Sumaira Abdullah, Senior Registrar, Islamabad Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMDC
Record Dates: First submitted 2019-05-27; First posted 2019-06-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Melasma
Keywords: melasma; hydroquinone; silymarin
MeSH Terms: conditions — Melanosis | interventions — hydroquinone; Silymarin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroquinone group (Active Comparator): Hydroquinone 4% cream Cream applied once daily at night on affected areas for 3 months.
  Interventions: Drug: Hydroquinone 4% Cream
- Silymarin group (Experimental): Silymarin 0.7% cream Cream applied twice daily on affecectec areas for 3 months.
  Interventions: Drug: silymarin 0.7% cream

INTERVENTIONS:
Drug: Hydroquinone 4% Cream — Hydroquinone is tyrosinase inhibitor and thus inhibits melanogenesis.
  Arms: Hydroquinone group
Drug: silymarin 0.7% cream — Silymarin is a plant derived flavonoid, extracted from fruits and seeds of milk thistle.
  Arms: Silymarin group

SUMMARY:
A randomized clinical trial will be done on 92 patients , randomly divided into two groups by lottery method to compare the efficacy and safety of topical silymarin cream 0.7% with topical 4% hydroquinone cream. Patients will be treated for 3 months and for the next 3 months will be followed up for relapse of melasma.

DETAILED DESCRIPTION:
A comparative study done by Nofal A et al, comparing the effectiveness and safety of topical silymarin versus hydroquinone, concluded that silymarin cream can be used as more potent and safer treatment option for the treatment of melasma.8 Two different concentrations of silymarin cream (0.7% and 1.4%) were used in this study and the results showed that both the groups have no statistically significant difference in terms of therapeutic response (mean of percentage reduction in MASI was 39.21 for 0.7% silymarin cream group and 33.84 for 1.4% silymarin cream group). Additionally relapse cases were identified in 7.14% of patients in both the groups. This shows that silymarin used at low concentration can prove to be more potent than at high concentration when it comes to effectiveness, cost and adverse effects. Therefore, I will compare 0.7% silymarin cream with 4% hydroquinone cream in my clinical trial for the treatment of melasma.

Rationale of this study is to observe the effects of this alternative treatment option and compare it with the first line drug so that it can be recommended in the guidelines as an alternative treatment option for melasma. The study by Nofal at al. was done in Egypt where most if the people have type 4 skin and environmental conditions are also similar to Pakistan. However a very small population group was included in the study. I want to do the same interventional trial on a larger population size to validate silymarin as an effective and safer treatment option.

Patients attending ANTH dermatology out patient, fulfilling the inclusion criteria will be inducted. Informed written consent will be taken from the enrolled patients and confidentiality will be maintained throughout the study. A detailed history will be taken focusing on duration and onset, family history, any relation to pregnancy, effect of exposure to sun, systemic inquiry and prior treatment sought. Fitzpatrick skin type and melisma pattern will be assessed. Melasma type will be assessed with the help of Wood's light examination. The severity of melasma will be assessed using MASI score. Random distribution of patients will be done through lottery method. Group A will be treated with topical hydroquinone 4% cream applied once daily at night and group B with silymarin 0.7% cream applied twice daily. All the patients will be advised to have proper sun protection measures, use physical protection like umbrella or a P cap and a wear sunscreen having a sun protective factor of at least 60. Patients will be advised not to use topical retinoids or any other product containing peroxide in it and not to apply the cream near eyes, mouth or nose. Patients will be asked to do a patch test on volar aspect of arms for 3 days before starting the treatment on face and immediately stop the treatment and report if she develops erythema and/or burning sensation with either drug. Digital photography will be taken at baseline and after every month during the treatment course till three months.

Patients will be booked for follow up at 1 month interval for 6 months. Treatment will be given for 3 months and will be followed up for the next 3 months (during which patients will be using only sun protection measures) to observe relapse of melasma. On follow up visits during treatment period, history will be taken regarding compliance to treatment and drug tolerance. The MASI score will be calculated at baseline and each follow up visit. Clinical efficacy will be assessed in terms of percent reduction in MASI score from baseline. Any adverse effect of treatment and patient's satisfaction using the short assessment of patient<s satisfaction will be measured at each visit. Information will be recorded on specially designed performas.

The data will be analyzed with the help of Statistical Package for Social Sciences (SPSS) version 25. Data will be presented as mean ± SD for quantitative variables (age, percent reduction of MASI, Short Assessment of Patient Satisfaction) and frequency with percentages for categorical variables (sun exposure, family history, previous therapy, melasma type, melasma pattern, melasma severity, burning and erythema). Independent sample t-test will be used to compare percent reduction in MASI score between both treatment groups at each follow up. Paired sample t-test will be used to compare the MASI score with baseline at each follow up visit within both groups. Chi-square test will be applied to compare the clinical efficacy, and safety in terms of any side effect between both groups throughout the study period. P-value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Female sex.
* Age 18 or older.
* Melasma of different severities, types and patterns

Exclusion Criteria:

* Pregnant or lactating females (Hydroquinone has pregnancy category C and it is not known if it is distributed in breast milk or not).
* Ongoing use of hormonal birth control pills or any hormonal therapy (as they cause hyperpigmentation).
* Use of topical anti melasma therapy within 3 months (efficacy of current therapy cannot be concluded).

  * Use of topical steroids within 3 months (as topical steroids will decrease hyperpigmentation).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Therapeutic response will be assessed in terms of percent reduction in MASI score from baseline to 1,2 and 3 month of treatment course and for next 3 months of follow up. | 6 months
  * >75% improvement as excellent
  * 50-75% improvement as good
  * 25-50% improvement as medium
  * < 25% improvement as poor

SECONDARY OUTCOMES:
b) Measurement of patient's satisfaction monthly for 6 months by the Short Assessment of Patient Satisfaction (SAPS). | 6 months
  * 0 - 10 very unsatisfied.
  * 11 - 18 unsatisfied.
  * 19 - 26 satisfied.
  * 27 - 28 very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Abdullah, MBBS, MCPS, MD, Principal Investigator — Senior Registrar in Dermatology
Locations (1):
- Islamabad medical and Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nofal A, Ibrahim AM, Nofal E, Gamal N, Osman S. Topical silymarin versus hydroquinone in the treatment of melasma: A comparative study. J Cosmet Dermatol. 2019 Feb;18(1):263-270. doi: 10.1111/jocd.12769. Epub 2018 Aug 26. PMID 30146802